CLINICAL TRIAL: NCT00819338
Title: The Effect of n-3 Polyunsaturated Fatty Acid Supplementation in Patients With Non-alcoholic Fatty Liver Disease
Brief Title: The Effect of n-3 Polyunsaturated Fatty Acid Supplements in Patients With Non-alcoholic Fatty Liver Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Richard Johnston, Doctor, University of Nottingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NottinghamNHST1; REC 08/H0403/14; R&D 08GA001
Record Dates: First submitted 2009-01-08; First posted 2009-01-09 (Estimated); Last update posted 2012-07-04 (Estimated); Status verified 2012-07

CONDITIONS: Non-alcoholic Fatty Liver Disease
Keywords: Non-alcoholic fatty liver disease; Polyunsaturated fatty acids; Omega-3
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- polyunsaturated (Active Comparator): 5g per day of polyunsaturated fatty acids (3.5g EPA and DHA).
  Interventions: Dietary Supplement: Efamax
- monounsaturated (Placebo Comparator): 5g a day of oleic enriched sunflower oil
  Interventions: Dietary Supplement: Efamax

INTERVENTIONS:
Dietary Supplement: Efamax — 5g daily as capsules for 3 months
  Other Names: oleic enriched sunflower oil

SUMMARY:
The principal purpose of this study is to determine whether increased intakes of n-3 polyunsaturated (omega-3) fatty acids will reduce the amount of fat stored in the liver in patients with non-alcoholic fatty liver disease.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) is present in 10-24% of the general adult population. The first step of NAFLD involves the accumulation of fat within the liver (steatosis). Steatosis occurs either due to defective generation, metabolism or excretion of fatty acids by the liver. The next step in NAFLD progression is inflammation, which commonly occurs due to pro-inflammatory stimuli. Persistent inflammation results in end-stage liver disease. NAFLD is associated with the metabolic syndrome, which is characterised by central obesity, insulin resistance, raised triglycerides and hypertension. With the current obesity epidemic, there is predicted to be greater numbers of patients with NAFLD in the future.

Polyunsaturated fatty acids (PUFAs) are essential components of our diet, though standard Western intakes are lower than the recommended amounts. Supplementing the long chain n-3 PUFAs (commonly termed omega-3), EPA and DHA, improves many of the metabolic syndrome features. They lower plasma triglycerides, and may improve insulin resistance.

The diet of NAFLD patients tends to be deficient in n-3 PUFAs and have an excessive intake of the harmful n-6 PUFAs. This pattern is mirrored in their liver lipid content as assessed at biopsy.

Currently there is no proven treatment for NAFLD. Animal studies and limited studies in patients have been supportive of a benefit with n-3 polyunsaturated fatty acids. This needs to be further assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 18 years
2. Liver biopsy diagnosis of NAFLD

Exclusion Criteria:

1. Excessive alcohol intake - > 21 units per week in men and > 14 in women
2. A further liver disease diagnosis
3. Poorly controlled diabetes - HbA1c > 8.0%, or use of insulin sensitisers
4. Pregnancy
5. Cirrhosis
6. Contraindications to MR scanning - pacemaker or metallic foreign body etc.
7. Changes in the dose or initiation of lipid altering medication within the preceding three months, such as statins, fibrates or systemic steroids
8. Use of n-3 PUFA supplements within the prior 4 months, an adequate washout period
9. Significant co-morbid inflammatory illnesses as determined by research team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2009-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Reduction of intrahepatic fat content as determined by magnetic resonance spectroscopy | 3 months

SECONDARY OUTCOMES:
Serum liver function tests, lipids, free fatty acids | 3 months
Insulin resistance as assessed by HOMA-IR and Adipose Tissue Insulin Resistance Index | 3 months
Liver saturated, monounsaturated and polyunsaturated fatty acid indexes as assessed by MR spectroscopy | 3 months
Visceral obesity as quantified by MRI, and the adipose derived serum leptin and adiponectin | 3 months
Primary assessment of the fibrotic and inflammatory status of the liver with serum TGF beta, TNF a, IL-6, IL-8, IL-8, IL-10 | 3 months
Further informative cytokine analyses: GM-CSF, IFN-G, IL-1B, IL-1RA, IL-2, IL-4, IL-5, MCP1 | 3 months
Compliance assessed by serum phospholipid fatty acids | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ian A Macdonald, PhD, Study Chair — Biomedical Sciences, University Hospital, Nottingham
Locations (1):
- Wolfson Digestive Diseases Centre, University Hospital, Nottingham, United Kingdom